CLINICAL TRIAL: NCT05481866
Title: Targeting Gut Microbiota and Metabolites for Very Preterm Infants Through Oropharyngeal Administration of Colostrum: Protocol for a Multicenter Randomized Controlled Trial
Brief Title: Targeting Gut Microbiota and Metabolites for Very Preterm Infants Through Oropharyngeal Administration of Colostrum
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Shenzhen People's Hospital (Other)
Collaborators: Shenzhen Bao'an Maternal and Child Health Hospital (Other); Longgang Maternal and Child Health Hospital, Shenzhen, Guangdong (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SZPH-2022-52
Record Dates: First submitted 2022-07-20; First posted 2022-08-01 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Gut Microbiota; Metabolites

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The intervention group will be given colostrum for oropharyngeal administration (Experimental): The intervention group will be given 0.2ml colostrum for oropharyngeal administration every 3 hours, which will start between the first 48 to 72 hours and continue for 5 consecutive days.
  Interventions: Other: Oropharyngeal administration of colostrum
- The control group will be given sterile water for oropharyngeal administration (Placebo Comparator): The control group will be given sterile water for oropharyngeal administration, and the administration scheme will be the same as above.
  Interventions: Other: Oropharyngeal administration of sterile water

INTERVENTIONS:
Other: Oropharyngeal administration of colostrum — The intervention group will be given 0.2ml colostrum for oropharyngeal administration every 3 hours.
  Arms: The intervention group will be given colostrum for oropharyngeal administration
Other: Oropharyngeal administration of sterile water — The control group will be given 0.2ml sterile water for oropharyngeal administration every 3 hours.
  Arms: The control group will be given sterile water for oropharyngeal administration

SUMMARY:
Background: Oropharyngeal administration of colostrum (OAC) has an immune stimulating effect on oropharyngeal-associated lymphoid tissue, and can also promote the maturation of the gastrointestinal tract. However, how OAC promotes intestinal maturation in preterm infants by altering the gut microbiota remains unclear. We aim to assess the changes of gut microbiota and metabolites after OAC in very preterm infants.

Methods: A multicenter, double-blind, randomized controlled trial will be conducted in 3 large NICUs in Shenzhen, China, for preterm infants with gestational age less than 32 weeks and birth weight less than 1500g. The intervention group will be given 0.2ml colostrum for oropharyngeal administration every 3 hours, which will start between the first 48 to 72 hours and continue for 5 consecutive days; The control group will be given sterile water for oropharyngeal administration, and the administration scheme will be the same as above. Stool samples will be collected at the first defecation and the 7th day after birth. It is estimated that 320 preterm infants will participate in the study within 1 year. 16sRNA gene sequencing and liquid chromatography-mass spectrometry will be used to analyze the effect of OAC on gut microbiota and metabolites.

Discussion: The proposal advocates for the promotion of OAC as a safe and relatively beneficial initiative among neonatal intensive care units, and this initiative may contribute to the establishment of a dominant intestinal flora. Findings of this study may help to improve the health outcomes of preterm infants by constructing targeted gut microbiota in future studies.

DETAILED DESCRIPTION:
Preterm infants with gestational age < 32 weeks and weight < 1500g will be evaluated. Infants who met the inclusion criteria will be randomly divided into two groups according to the ratio of 1:1. The intervention group will be given oropharyngeal colostrum every 3 hours for 5 days; the control group will be given sterile water with the same dosage and administration scheme. Stool samples will be collected at the first defecation and the 7th day to detect the gut microbiota and metabolites.

ELIGIBILITY:
Inclusion criteria:

* gestational age less than 32 weeks and birth weight less than 1500g;
* admission to NICU ≤ 24 hours;
* be able to start the agreement within 72 hours of birth.

Exclusion criteria:

* birth asphyxia (defined as umbilical artery / first hour arterial PH < 7.0 or cardiopulmonary resuscitation in the delivery room);
* birth complicated with severe gastrointestinal malformations (such as intestinal atresia, esophago-tracheal fistula, intestinal rotation abnormalities, congenital megacolon);
* prenatal diagnosis of congenital chromosomal abnormalities or suspected congenital genetic metabolic diseases;
* maternal drug abuse or contraindications to breastfeeding (HIV and cytomegalovirus infection).

Max Age: 32 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 320 (Estimated)
Dates: Start 2022-10 (Estimated); Primary Completion 2023-10 (Estimated); Study Completion 2023-10 (Estimated)

PRIMARY OUTCOMES:
A between-group difference in gut microbial alpha diversity will be measured by Shannon diversity index at the 7th day. | 1 year
  Shannon diversity Index explains species richness and evenness, which is one of the alpha diversity indexes and less affected by rare species.
Between-group differences in the concentration of fecal metabolites (short chain fatty acids) will be quantitatively measured by non targeted liquid chromatography-mass spectrometry (LC-MS) at the 7th day. | 1 year
  Non-targeted LC-MS will be used to evaluate short chain fatty acids and other organic acids and alcohols. The relative and absolute quantitative results of metabolites will be calculated by fold change (FC) value, and the difference of metabolite expression between the two groups will be explored.

SECONDARY OUTCOMES:
A between-group difference in the Simpson diversity index at the 7th day | 1 year
  Simpson diversity index explains species richness, which is one of the alpha diversity indexes and susceptible to rare species.
A between-group difference in the Chao1 diversity index at the 7th day. | 1 year
  Chao1 diversity index explains species richness, which is one of the alpha diversity indexes.
Proportion of gut microbiota (phylum and genus level）at the 7th day. | 1 year
  After preprocessing to remove low-quality sequences, the original data will be analyzed according to the steps of 16S rRNA discovery, clustering and identification. Calculate the number of operational taxonomic units (OTUs) of each sample at a 97% sequence similarity level. A specific taxonomic units represents a specific species.
Gut microbial beta diversity explaining between-sample dissimilarity will be calculated using the Vegan package. | 1 year
  Adonis permutational multivariate analysis of variance of Bray-Curtis distances with 9999 permutations will be used to compare the microbial community structure between each of the two groups at the 7th day.
Correlation between dominant microbiota and metabolites | 1 year
  The correlation between the relative abundance of dominant bacterial taxa from 16S rRNA gene sequencing and the intensity of metabolites of interest will be determined by sparse partial least squares regression (SPLs) at the first defecation at the 7th day.

CONTACTS AND LOCATIONS:
Overall Officials: Zhangbin Yu, PhD, Principal Investigator — Shenzhen People's Hospital
Locations (1):
- Shenzhen People's Hospital, Shenzhen, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wang N, Zhang J, Yu Z, Yan X, Zhang L, Peng H, Chen C, Li R. Oropharyngeal administration of colostrum targeting gut microbiota and metabolites in very preterm infants: protocol for a multicenter randomized controlled trial. BMC Pediatr. 2023 Oct 16;23(1):508. doi: 10.1186/s12887-023-04346-x. PMID 37845612